CLINICAL TRIAL: NCT05867394
Title: The Effect of Stress Ball Application Before Coronary Angiography on Stress, Anxiety and Vital Signs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aysel Sesci (Other)
Responsible Party: Sponsor-Investigator, Aysel Sesci, principal investigator, Aksaray University
Organization: Aksaray University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Aksaray Üniversitesi
Record Dates: First submitted 2023-02-28; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Coronary Artery Disease
Keywords: coronary angiography; stress; anxiety; vital signs
MeSH Terms: conditions — Coronary Artery Disease; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Prospective Randomized Controlled Clinical Trial
Who Masked: Participant
Masking Description: Participants do not know which group they are in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress ball (Experimental): Data were collected by the investigator 25-30 minutes before coronary angiography and the first measurement of vital signs was made. After the stress ball application, State Anxiety Inventory data were collected for the second time and the second measurement of vital signs was made. Vital signs were measured and noted for the third time after coronary angiography.
  Interventions: Other: Stress ball
- Control (No Intervention): 25-30 minutes before the coronary angiography procedure, data were collected from the patients by the investigator and the first measurements of their vital signs were recorded. Vital signs were measured a second time just before coronary angiography without any intervention. Vital signs were measured and recorded for the third time after coronary angiography ischemia.

INTERVENTIONS:
Other: Stress ball — Stress ball squeeze
  Arms: Stress ball

SUMMARY:
It aimed to examine stress, anxiety and resorting to life paths to enable researchers to contain this stress.

DETAILED DESCRIPTION:
Stress and anxiety lives of patients before coronary angiography. The stress and anxiety they experience also affect their vital signs. The researchers aimed to examine the ways the stress ball affected their patients' stress, anxiety, and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over
* For those who will undergo coronary angiography for the first time
* Able to read and write
* Not diagnosed with anxiety disorder and not using medication for it
* No physical disability to use the stress ball
* Cognitive health levels consist of individuals who are suitable for answering data collection forms.

Exclusion Criteria:

* Unconscious and not fully oriented
* Sight and hearing problems
* Alzheimer's disease and other types of dementia
* Having a severe psychiatric problem that cannot answer the questions
* Those who came with MI (myocardial infarction) and performed CAG
* Individuals who are closed to communicating are not included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
State Anxiety Score | Change in state anxiety score within one day
  Scale measuring patients' anxiety. The scores obtained from the scale vary between 20 and 80. A large score indicates high anxiety, and a small score indicates low anxiety.

SECONDARY OUTCOMES:
Distress Thermometer | Only on day 1, 2 times a day (same day).
  It is a scale that measures the patient's stress level. The scale is scored between 0 and 10 points. A score of 0 indicates no stress, and a score of 10 indicates extreme stress.
Systolic Blood Pressure Value (mmHg) | Only on day 1, 2 times a day (same day).
  The effect of the intervention on systolic blood pressure is examined.
Diastolic Blood Pressure Value (mmHg) | It will be measured 3 times a day (same day) on day 1 only.
  The effect of the intervention on diastolic blood pressure is examined.
Heart Rate/Minute Value | It will be measured 3 times a day (same day) on day 1 only.
  The effect of the intervention on the heart rate is examined.
Respiratory Rate/Minute Value | It will be measured 3 times a day (same day) on day 1 only.
  The effect of the intervention on the respiratory rate is examined.
Peripheral Oxygen Saturation (SpO2) Value | It will be measured 3 times a day (same day) on day 1 only.
  The effect of the intervention on peripheral oxygen saturation is examined.

CONTACTS AND LOCATIONS:
Locations (1):
- Aysel SESCİ, Aksaray, University, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Study protocol